CLINICAL TRIAL: NCT00902291
Title: A Global, Multi-center, Open-label, Phase 2 Study of AGS-1C4D4 Given in Combination With Gemcitabine in Subjects With Metastatic Pancreatic Cancer
Brief Title: A Study of AGS-1C4D4 Given in Combination With Gemcitabine in Subjects With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Agensys, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008002; 2009-009194-99 (EudraCT Number)
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-08

CONDITIONS: Carcinoma, Pancreatic Ductal; Pancreatic Cancer; Pancreatic Disease
Keywords: Clinical Trial, Phase II; Combination Drug Therapy; Gemcitabine; AGS-1C4D4; Pancreatic Cancer
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal; Pancreatic Neoplasms; Pancreatic Diseases | interventions — MK-4721; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Gemcitabine monotherapy (Active Comparator)
  Interventions: Biological: Gemcitabine
- 2. Gemcitabine plus AGS-1C4D4 (Experimental)
  Interventions: Biological: AGS-1C4D4; Biological: Gemcitabine

INTERVENTIONS:
Biological: AGS-1C4D4 — IV infusion
  Arms: 2. Gemcitabine plus AGS-1C4D4
Biological: Gemcitabine — IV infusion

SUMMARY:
A study to evaluate AGS-1C4D4 administered in combination with Gemcitabine chemotherapy in subjects with Metastatic Pancreatic Cancer.

DETAILED DESCRIPTION:
A disease assessment will be performed at study week 8 (± 3 days) by the investigator. The assessment will be based both on changes in clinical symptoms, and radiographic images. Subjects without evidence of disease progression may continue to receive treatment based on their original treatment assignment until disease progression or intolerability. Disease assessments will be performed every 8 weeks during the extended period. A safety follow-up visit will occur 4 weeks after the last dose infusion of AGS-1C4D4 and/or gemcitabine.

Post-Treatment: Subjects terminating from protocol therapy for reasons unrelated to documented disease progression will be followed by telephone contact every 2 months until they begin a new anticancer therapy, their disease progresses, they die, become lost to follow-up or withdrawal consent for further follow-up, whichever of these events occurs first.

Overall survival: All subjects will be followed by telephone contact every 2 months until death, loss to follow-up, or withdrawal of consent, whichever of these events occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed metastatic adenocarcinoma of the pancreas (AJCC Stage IV). Subjects with islet cell neoplasms are excluded
* Non-measurable or measurable disease based on the RECIST criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Life expectancy of > 3 months
* Hematologic function, as follows:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Hemoglobin ≥ 9 g/dL (transfusion independent)
* Renal function, as follows:

  * Creatinine ≤ 2.0 mg/dL
* Hepatic function, as follows:

  * Aspartate aminotransferase (AST) ≤ 2.5 x ULN or ≤ 5 x ULN if known liver metastases.
  * Alanine aminotransferase (ALT) ≤ 2.5 x ULN or ≤ 5 x ULN if known liver metastases
  * Bilirubin ≤ 2 x ULN
* INR < 1.3 (or ≤ 3 if on warfarin for therapeutic anti-coagulation)

Exclusion Criteria:

* Prior systemic therapy for metastatic pancreatic cancer

  * Subjects who have received adjuvant treatment with gemcitabine and who had relapse metastatically are allowed
  * Subjects with advanced local disease who have received treatment with gemcitabine and in whom progression has been observed with the onset of metastases less than 6 months are excluded
* Chemotherapy and/or radiation within 4 weeks of study enrollment
* Prior monoclonal antibody therapy within 60 days of study enrollment
* Known brain or leptomeningeal disease
* History of other primary malignancy, unless:

  * Curatively resected non-melanomatous skin cancer
  * Other malignancy curatively treated with no known active disease present and no treatment administered for the last 3 years
* Active angina or Class III or IV Congestive Heart Failure (New York Heart Association CHF Functional Classification System)
* Use of any investigational product within 4 weeks of study enrollment
* Major surgery (that requires general anesthesia) within 4 weeks before study enrollment
* Women who are pregnant (confirmed by positive pregnancy test) or lactating
* Man or woman of childbearing potential not consenting to use adequate contraceptive precautions during the course of the study and for 4 weeks after the last AGS-1C4D4 and/or gemcitabine infusion administration
* Subject known to be human immunodeficiency, hepatitis B or hepatitis C virus positive
* Active serious infection not controlled with antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2009-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Survival rate at 6 months | 6 months

SECONDARY OUTCOMES:
Overall Survival (OS) | Throughout treatment period and post-treatment every 2 months until death, or subject discontinues the study
Progression free survival (PFS) | Throughout treatment period or post-treatment every 2 months until disease progression or death, respectively, or subject discontinues the study
Change in level of serum tumor marker CA 19-9 | Week 1, Week 4, Week 7 and every 3 weeks during the extended treatment period
Incidence of anti-AGS-1C4D4 antibody formation | Week 1, Week 7 and every 8 weeks during the extended treatment period
Objective Response Rate (Partial Response or better per RECIST criteria version 1.1 | Week 8, and every 8 weeks during the extended treatment period
Disease Control (Stable Disease or better per RECIST criteria) | Week 8, and every 8 weeks during the extended treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Agensys, Inc.
Locations (36):
- United States (15):
  - University of California San Diego Medical Center, La Jolla, California
  - Palm Beach Institute of Hematology and Oncology, Boynton Beach, Florida
  - University of Miami, Miami, Florida
  - Medical Oncology LLC, Baton Rouge, Louisiana
  - Annapolis Oncology Center, Annapolis, Maryland
  - Dana Farber Cancer Center, Boston, Massachusetts
  - Virginia G. Piper Cancer Center, Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Regional Oncology Center, Syracuse, New York
  - Kaiser Permanente Northwest Region Oncology Hematology, Portland, Oregon
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Baptist Regional Cancer Center, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Div. of Medical Oncology, Nashville, Tennessee
  - Alan B. Pearson Regional Cancer Center Lynchburg Hematology Oncology Clinic, Lynchburg, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- France (6):
  - Chu Estaing, Clermont-Ferrand
  - Centre Jean Bernard, Oncologie médicale, Le Mans
  - Centre Régional de Lutte Contre le Cancer-Centre Oscar Lambret, Lille
  - Hôpital du Haut Lèvêque, Service d'Hepato Gastroentérologie, Pessac
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Hôpital Charles Nicolle, Rouen
- Russia (9):
  - State Institution of Healthcare "Arkhangelsk Regional Clinical Oncology Dispensary", Arkhangelsk
  - Regional Oncology Dispensary, Ivanovo
  - Clinical Oncology Dispensary of Republic of Tatarstan, Kazan'
  - State Healthcare Institution "Leningrad Regional Oncologic Dispensary", Kuzmolovo
  - Non-state Healthcare Institution N.A. Semashko Central Clinical Hospital #2 of JSC "Russian Railway", Moscow
  - Medical Radiology Research Center of Russian Medical Academy, Obninsk
  - State Healthcare Institution of Omsk Region "Clinical Oncologic Dispensary", Omsk
  - Saint Petersburg State Healthcare Institution "Municipal Clinical Oncology Dispensary", Saint Petersburg
  - State Educational Institution "S.M. Kirov Military Medical Academy of Ministry of Defense of Russia", Saint Petersburg
- Spain (3):
  - Hospital Clinic i Provincial de Barcelona, Servicio de Oncologia, Barcelona
  - Madrid
  - Hospital Virgen de la Salud, Servicio Oncologia, Toledo

REFERENCES:
- [Background] Wolpin BM, O'Reilly EM, Ko YJ, Blaszkowsky LS, Rarick M, Rocha-Lima CM, Ritch P, Chan E, Spratlin J, Macarulla T, McWhirter E, Pezet D, Lichinitser M, Roman L, Hartford A, Morrison K, Jackson L, Vincent M, Reyno L, Hidalgo M. Global, multicenter, randomized, phase II trial of gemcitabine and gemcitabine plus AGS-1C4D4 in patients with previously untreated, metastatic pancreatic cancer. Ann Oncol. 2013 Jul;24(7):1792-1801. doi: 10.1093/annonc/mdt066. Epub 2013 Feb 28. PMID 23448807